CLINICAL TRIAL: NCT05907564
Title: Evaluate the Safety and Efficacy of the Aventus Thrombectomy System for Aspiration Thrombectomy in Subjects With Acute Pulmonary Embolism
Brief Title: Aventus Thrombectomy System Pulmonary Embolism Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inquis Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-0001
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Embolism; Embolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Lung Diseases; Respiratory Tract Diseases
Keywords: Pulmonary Embolism; Clot; Thromboembolism; Thrombectomy; Right Heart Strain
MeSH Terms: conditions — Pulmonary Embolism; Embolism; Embolism and Thrombosis; Vascular Diseases; Cardiovascular Diseases; Lung Diseases; Respiratory Tract Diseases; Thromboembolism | interventions — Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Experimental): Device: Aventus Thrombectomy System
  Interventions: Device: Thrombectomy

INTERVENTIONS:
Device: Thrombectomy — Use of Aventus Thrombectomy System to treat pulmonary embolism

SUMMARY:
Evaluate the safety and efficacy of the Aventus Thrombectomy System for aspiration thrombectomy in subjects with acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years
2. Subject or legally authorized representative (LAR) is willing and able to provide written informed consent prior to receiving any non-standard of care protocol specific procedures
3. Subject is willing and able to comply with all protocol required follow-up visits
4. PE symptom(s) duration ≤ 14 days from index procedure
5. PE diagnosis ≤ 48 hours prior to index procedure
6. CTA evidence of proximal PE (filling defect in at least one main or lobar pulmonary artery based on Investigator determination)
7. CTA evidence of dilated RV with an RV/LV ratio of ≥ 0.9 at baseline based on Investigator determination
8. Systolic blood pressure ≥ 90 mmHg without need for vasopressors (initial SBP may be ≥ 80 mmHg if the pressure recovers to ≥ 90 mmHg with intravenous fluids prior to index procedure)
9. Stable heart rate < 130 BPM prior to index procedure
10. Subject is deemed medically eligible for interventional procedure(s), per institutional guidelines and clinical judgment

Exclusion Criteria:

1. Prior PE ≤ 180 days from index procedure
2. Current hospitalization for other condition(s)
3. Thrombolytic use ≤ 14 days of baseline CTA
4. Pulmonary hypertension with peak pulmonary artery systolic pressure > 70 mmHg by right heart catheterization
5. FiO2 requirement > 40% or > 6 LPM to keep oxygen saturation > 90%
6. Hematocrit < 28% within 6 hours of index procedure
7. Platelets < 100,000/μL
8. Serum creatinine > 1.8 mg/dL
9. International normalized ratio (INR) > 3
10. Presence of intracardiac lead in the right ventricle or right atrium placed < 180 days prior to index procedure
11. Cardiovascular or pulmonary surgery ≤ 7 days prior to index procedure
12. Actively progressing cancer treated by chemotherapeutics
13. Known bleeding diathesis or coagulation disorder
14. Left bundle branch block
15. History of severe or chronic pulmonary arterial hypertension
16. History of chronic left heart disease with left ventricular ejection fraction ≤ 30%
17. History of uncompensated heart failure
18. History of underlying lung disease that is oxygen dependent
19. History of chest irradiation
20. History of heparin-induced thrombocytopenia (HIT)
21. Any contraindication to systemic or therapeutic doses of heparin or anticoagulants
22. Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
23. Imaging evidence or other evidence that suggests, in the opinion of the Investigator, the Subject is not appropriate for aspiration thrombectomy intervention such as the inability to navigate to target location, predominantly chronic clot or non-clot embolus
24. Life expectancy of < 90 days, as determined by Investigator
25. Female who is pregnant or nursing
26. Current participation in another investigational drug or device treatment study that has not reached the primary endpoint or the Investigator feels would impact their ability to participate in this clinical trial
27. Subject has known residual Iliac Deep Vein Thrombosis (DVT), Inferior Vena Cava (IVC) clot or clot in transit (right atrium and/or right ventricular)
28. Subject on extracorporeal membrane oxygenation (ECMO)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in RV/LV Ratio | From Baseline to 48 hours
  Change in RV/LV Ratio per CTA
Major Adverse Event Rate | From Index Procedure to 48 hours
  Composite of device related MAEs including death, major bleed, clinical deterioration, pulmonary vascular injury, and cardiac injury

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Principal Investigator — University Hospitals; Saher Sabri, MD, Principal Investigator — MedStar Health
Locations (26):
- United States (26):
  - Honor Health, Scottsdale, Arizona
  - NorthBay Medical Center, Fairfield, California
  - MemorialCare, Long Beach, California
  - El Camino Health, Mountain View, California
  - Sutter Health, Sacramento, California
  - Hartford Hospital, Hartford, Connecticut
  - Medstar, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Ascension St. Vincent, Indianapolis, Indiana
  - Ochsner Health, New Orleans, Louisiana
  - McLaren Health Care, Bay City, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Providence, Southfield, Michigan
  - CentraCare Heart and Vascular, Saint Cloud, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - University Hospitals, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - ProMedica - Jobst Vascular, Toledo, Ohio
  - Ascension St. John, Tulsa, Oklahoma
  - The Miriam Hospital, Providence, Rhode Island
  - Centennial Medical Center (HCA), Nashville, Tennessee
  - Ascension Seton, Austin, Texas

IPD SHARING:
Plan to Share IPD: No